CLINICAL TRIAL: NCT05101434
Title: Gingivitis and Periodontitis as a Risk Factor for Stroke
Status: Completed | Type: Observational
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, Muhammad Hassan, Registrar Neurology, Shaheed Zulfiqar Ali Bhutto Medical University
Other Study IDs: Gingivitis and Stroke
Record Dates: First submitted 2021-10-18; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Gingivitis; Periodontitis; Stroke
MeSH Terms: conditions — Gingivitis; Periodontitis; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Periodontal Probing — with the help Michigan probe, periodontal pocket measurement was done.
  Other Names: ROAG revised oral assessment guide; Community periodontal index; Gingival Index

SUMMARY:
Periodontitis and gingivitis are one of the most infectious diseases in humans. Several studies have been carried out on the dependence of periodontitis and stroke. The aim of this study was to investigate gingivitis and periodontitis as risk factors for stroke in the Pakistani population.

DETAILED DESCRIPTION:
Epidemiologic studies have shown that cerebrovascular accident (CVA) is the 3rd cause of death in developed countries with 0.8 % prevalence in the whole population. Although, the prevalence rate of stroke is reduced yet is one of the most important health problems in the United State. Periodontitis and gingivitis are the two most infectious man diseases. Today, it is estimated that about 35% of people over 30-year-old in America and 50-55% of people in developing countries are involved with these diseases.

These diseases are due to the practice of chronic bacterial infection and the inflammatory response of the host. The relationship between periodontitis and CVA was first introduced by Mackenzi and Millard in 1963 but the importance of this issue was not understood. Periodontal infection can be a complex multiphase disease by associating this infection with organ systems such as cardiovascular, endocrine, reproductive, and respiratory systems. Nowadays, periodontitis is considered a risk factor for atherosclerosis and thromboembolic disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed stroke by using brain imaging from magnetic resonance imaging and/or computerized tomography.

Exclusion Criteria:

* Not willing to participate
* Neurological complications other than stroke

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients with stroke (both ischemic and hemorrhagic)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Gingivitis | baseline
  Measurement of bleeding site while probing and this was done with gingival index
Periodonitis | baseline
  Measurement of periodontal pockets while probing and this was done with community periodontal idex

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hassan, MD, Principal Investigator — Shaheed Zulfiqar Ali Bhutto Medical University
Locations (1):
- Shaheed Zulfiqar Ali Bhutto Medical University, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared on reasonable demand